CLINICAL TRIAL: NCT01676051
Title: Efficacy of Surgical Preparation Solutions in Hand Surgery
Brief Title: Surgical Prep in Hand Surgery
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John Fowler, Fellow, University of Pittsburgh
Other Study IDs: PRO12080340
Record Dates: First submitted 2012-08-23; First posted 2012-08-30 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Surgical Scrubbing; Disinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Chloraprep
  Interventions: Other: Skin culture
- Duraprep
  Interventions: Other: Skin culture
- Betadine only
  Interventions: Other: Skin culture

INTERVENTIONS:
Other: Skin culture — Culture swab used to culture skin adjacent to incision

SUMMARY:
The purposes of this study are to identify the common bacterial flora on the hand and evaluate the efficacy of readily available skin-preparation solutions in the elimination of bacterial pathogens from the surgical site following skin preparation. The null hypothesis is that there is no difference in the efficacy of Chloraprep, Duraprep, and betadine in pre-operative skin preparation in clean, elective hand surgery cases.

ELIGIBILITY:
Inclusion Criteria:

* the following procedures (carpal tunnel release, trigger finger release, cyst excision, 1st dorsal compartment release)

Exclusion Criteria:

* prisoners
* pregnant women

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing clean, elective hand surgery without implants
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of positive cultures | after skin prep solution has dried

CONTACTS AND LOCATIONS:
Overall Officials: John Fowler, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Montefiore Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Savage JW, Weatherford BM, Sugrue PA, Nolden MT, Liu JC, Song JK, Haak MH. Efficacy of surgical preparation solutions in lumbar spine surgery. J Bone Joint Surg Am. 2012 Mar 21;94(6):490-4. doi: 10.2106/JBJS.K.00471. PMID 22437997
- [Background] Saltzman MD, Nuber GW, Gryzlo SM, Marecek GS, Koh JL. Efficacy of surgical preparation solutions in shoulder surgery. J Bone Joint Surg Am. 2009 Aug;91(8):1949-53. doi: 10.2106/JBJS.H.00768. PMID 19651954
- [Background] Ostrander RV, Botte MJ, Brage ME. Efficacy of surgical preparation solutions in foot and ankle surgery. J Bone Joint Surg Am. 2005 May;87(5):980-5. doi: 10.2106/JBJS.D.01977. PMID 15866959